CLINICAL TRIAL: NCT01134107
Title: A Double-Blind, Randomized, Crossover Trial of CSII Reservoir In-use Comparing Insulin Lispro Formulation to Insulin Aspart in Patients With Type 1 Diabetes Mellitus
Brief Title: Insulin Lispro 6 Days Versus Insulin Aspart 6 Days in Pump Use
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 12175; F3Z-MC-IOPW (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro 6 Day (6D) (Experimental)
  Interventions: Drug: Insulin Lispro 6 Day (6D)
- Insulin Aspart 6 Day (6D) (Active Comparator)
  Interventions: Drug: Insulin Aspart 6 Day (6D)

INTERVENTIONS:
Drug: Insulin Lispro 6 Day (6D) — Administered by infusion pump for 12 week treatment period
  Other Names: Insulin Lispro Formulation; Humalog; LY275585
  Arms: Insulin Lispro 6 Day (6D)
Drug: Insulin Aspart 6 Day (6D) — Administered by infusion pump for 12 week treatment period
  Arms: Insulin Aspart 6 Day (6D)

SUMMARY:
Patients will continue to use their current insulin pump for this study. Patients will receive insulin lispro and insulin aspart during this study. One medication will be taken for 12 weeks and then the other medication for 12 weeks. Neither the patient nor the study doctor will know which medication is being taken at any time. The order in which the two medications are taken will be determined by chance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes (World Health Organization criteria) for at least 24 months
* Treated with continuous subcutaneous insulin infusion (CSII) therapy for the previous 6 months
* Mean total daily insulin dose for 3 days prior to screening less than or equal to 46 units/day if using a 300-Unit reservoir, less than or equal to 30 units/day if using a 200 unit reservoir, or less than or equal to 26 units/day if using a 180 unit reservoir
* Baseline body mass index (BMI) less than or equal to 35.0 kilograms per meter squared (kg/m2)
* Baseline glycated hemoglobin A1c (HbA1c) 5% to 9%

Exclusion Criteria:

* Impaired renal function (serum creatinine greater than or equal to 2.0 milligrams per deciliter (mg/dL))
* Legal blindness
* Have had any episode in the 12 months prior to screening of hypoglycemic coma, seizures, or disorientation
* Have had hypoglycemia unawareness (routinely asymptomatic at blood glucose less than 45 mg/dL [2.5 millimoles per liter (mmol/L)]) in the 12 months prior to screening.
* Have had any emergency room visits or hospitalizations due to poor glucose control in the 12 months prior to screening.
* Have had a pump-related infusion site abscess in the 12 months prior to screening.
* Have had multiple, clinically significant occlusions as judged by the investigator.
* Have had any infection with Staphylococcus aureus in the past 5 years
* Have one of the following concomitant diseases: presence of clinically significant hematologic, oncologic, renal, cardiac, hepatic, or gastrointestinal disease, or any other serious disease considered by the investigator to be exclusionary.
* Participants with malignancy other than basal cell or squamous cell skin cancer who have not yet been treated, are currently being treated, or who were diagnosed less than 5 years ago.
* Have had a blood transfusion or severe blood loss within the 3 months prior to screening or have known hemoglobinopathy, hemolytic or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with HbA1c methodology.
* Are receiving chronic systemic glucocorticoid therapy, or have received such therapy within the 4 weeks preceding screening.
* Have an irregular sleep/wake cycle in the investigator's opinion.
* Have a known hypersensitivity or allergy to any of the study insulins or their excipients
* Are breastfeeding or pregnant, or intend to become pregnant during the course of the study, or are sexually active women of childbearing potential not actively practicing birth control by a method determined by the investigator to be medically acceptable.
* Are currently enrolled in, or discontinued within the last 30 days from a clinical trial involving off-label use of an investigational drug or device, or currently enrolled in any other type of medical research not to be scientifically or medically compatible with this study.
* Are unwilling or unable to comply with the use of a data collection device to directly record data from the participant.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corbeil-Essonnes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Rochelle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Narbonne
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludwigshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuwied
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Potsdam
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Békéscsaba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nyíregyháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zalaegerszeg

RESULTS

PARTICIPANT FLOW:
Groups:
- Lispro 6D/Aspart 6D: Insulin Lispro 6 Day (6D) administered by infusion pump for 12 weeks, followed by Insulin Aspart 6D administered by infusion pump for 12 weeks.
- Aspart 6D/Lispro 6D: Insulin Aspart 6D administered by infusion pump for 12 weeks, followed by Insulin Lispro 6D administered by infusion pump for 12 weeks.
Period: Period 1-First Treatment Intervention
Arm/Group | Lispro 6D/Aspart 6D | Aspart 6D/Lispro 6D
Started | 67 | 66
Received at Least One Dose of Study Drug | 66 | 66
Completed | 61 | 61
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Entry Criteria Not Met | 1 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Physician Decision | 1 | 0
Period: Period 2-Second Treatment Intervention
Arm/Group | Lispro 6D/Aspart 6D | Aspart 6D/Lispro 6D
Started | 61 | 61
Completed | 57 | 61
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lispro 6D/Aspart 6D: Insulin Lispro 6D administered by infusion pump for 12 weeks, followed by Insulin Aspart 6D administered by infusion pump for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Lispro 6D/Aspart 6D | Aspart 6D/Lispro 6D | Total
Number analyzed (Participants) | 67 | 66 | 133
Age Continuous [Mean (Standard Deviation); unit: years] | 40.71 (11.91) | 44.73 (12.96) | 42.70 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 45 | 93
  Male | 19 | 21 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  White | 67 | 66 | 133
Region of Enrollment [Number; unit: participants]
  France | 15 | 14 | 29
  Hungary | 33 | 37 | 70
  Germany | 19 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean of Last Six 7-point Self Monitored Blood Glucose (SMBG) Taken on Day 6 for Insulin Lispro 6D and Insulin Aspart 6D Pump Reservoir In-use
Time Frame: Day 6 of each reservoir cycle for the last 6 weeks of each 12-week treatment period (Week 7 through Week 12)
Population: All randomized participants who completed at least one post-randomization visit. Those included in the primary analysis had to have at least one reservoir in-use cycle with an SMBG measurement on Day 6 during the pre-specified collection period.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Groups:
- Insulin Lispro 6D: Insulin Lispro 6D administered by infusion pump for 12 week treatment period
- Insulin Aspart 6D: Insulin Aspart 6D administered by infusion pump for 12 week treatment period
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 118 | 118
millimoles per liter (mmol/L) | 8.83 (1.55) | 8.43 (1.97)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; This was the primary gated analysis; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 0.6 mmol/L was used; Least Squares Mean Difference = 0.36, 95% CI 2-sided [0.06 to 0.66] — Least Squares Mean Difference = Insulin Lispro 6 Day minus Insulin Aspart 6 Day; adjusted for Treatment + Sequence + Period + Baseline HbA1c

2. Secondary Outcome: Mean SMBG
Description: Mean SMBG for combined periods; all reported SMBG values on Days 1-6, Day 2, and Day 6 for Insulin Lispro 6D and Insulin Aspart 6D.
Time Frame: Days 1-6 and Day 2 and Day 6 for each reservoir cycle throughout each 12-week treatment period
Population: All randomized participants who completed at least one post-randomization visit and one SMBG measurement on a Day 6, or Day 2 depending on the analysis, for the respective treatment arm: insulin lispro 6D and insulin aspart 6D.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 126 | 126
millimoles per liter (mmol/L)
  SMBG Days 1-6 (N=124, 124) | 8.70 (2.51) | 8.47 (2.46)
  SMBG Day 2 | 8.56 (2.51) | 8.40 (2.47)
  SMBG Day 6 (N=124, 124) | 8.93 (2.68) | 8.57 (2.64)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 0.6 mmol/L was used; Least Squares Mean Difference = 0.18, 95% CI 2-sided [-0.10 to 0.47] — Least Squares Mean Difference = Insulin Lispro 6 Day (Day 1-6) minus Insulin Aspart 6 Day (Day 1-6); adjusted for Treatment + Sequence + Period + Baseline HbA1c
Statistical Analysis 2: Comparison: Insulin Lispro 6D; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 0.6 mmol/L was used; Least Squares Mean Difference = 0.42, 95% CI 2-sided [0.25 to 0.58] — Least Squares Mean Difference = Insulin Lispro 6 Day (Day 6) minus Insulin Lispro 6 Day (Day 2); adjusted for DayGroup + Period + Baseline HbA1c

3. Secondary Outcome: Mean Daily Insulin Dose (Total, Basal, and Bolus)
Time Frame: Days 1-6 for each reservoir cycle throughout each 12-week treatment period
Population: All randomized participants who completed at least one post-randomization visit. Participants included in insulin analyses are only those for whom data existed regarding insulin dose.
Measure: Mean (Standard Deviation); unit: Units (U) of insulin
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 119 | 119
Units (U) of insulin
  Daily Total Insulin | 32.90 (8.43) | 32.48 (8.42)
  Daily Basal Insulin | 17.83 (5.26) | 17.71 (5.27)
  Daily Bolus Insulin (N=116, 117) | 16.26 (6.21) | 16.09 (6.23)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; Least Squares Mean Difference = 0.38, 95% CI 2-sided [-0.13 to 0.88] — Daily Total Insulin: Least Squares Mean Difference = Insulin Lispro 6 Day minus Insulin Aspart 6 Day; adjusted for Treatment + Sequence + Period + Baseline Insulin Basal/Bolus/Total Dose
Statistical Analysis 2: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; Least Squares Mean Difference = 0.02, 95% CI 2-sided [-0.26 to 0.31] — Daily Basal Insulin: Least Squares Mean Difference = Insulin Lispro 6 Day minus Insulin Aspart 6 Day; adjusted for Treatment + Sequence + Period + Baseline Insulin Basal/Bolus/Total Dose
Statistical Analysis 3: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; Least Squares Mean Difference = 0.23, 95% CI 2-sided [-0.15 to 0.60] — Daily Bolus Insulin: Least Squares Mean Difference = Insulin Lispro 6 Day minus Insulin Aspart 6 Day; adjusted for Treatment + Sequence + Period + Baseline Insulin Basal/Bolus/Total Dose

4. Secondary Outcome: Change From Baseline to 12 Weeks for Each Treatment in Glycated Hemoglobin A1c (HbA1c) Values
Time Frame: Baseline, endpoint for each 12-week treatment period
Population: All randomized participants who completed at least one post-randomization visit, and had a baseline and a post-randomization HbA1c measurement for the respective treatment period. Last Observation Carried Forward (LOCF) method was utilized in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 127 | 126
percentage of HbA1c | -0.16 (0.54) | -0.31 (0.50)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; Least Squares Mean Difference = 0.16, 95% CI 2-sided [0.08 to 0.24] — Least Squares Mean Difference = Insulin Lispro 6 Day minus Insulin Aspart 6 Day; adjusted for Treatment + Period + Sequence + Baseline HbA1c

5. Secondary Outcome: Number of Participants Who Achieve or Maintain a Glycated Hemoglobin A1c (HbA1c) Less Than or Equal to 6.5% and Less Than 7%
Time Frame: Endpoint for each 12-week treatment period
Population: All randomized participants who completed a post-randomization visit and had an HbA1c measurement for the respective treatment period.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 127 | 126
participants
  HbA1c ≤6.5% | 18 | 21
  HbA1c <7% | 38 | 56
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.39 to 1.63] — Odds Ratio of HbA1c ≤6.5% for Insulin Lispro 6 Day versus Insulin Aspart 6 Day
Statistical Analysis 2: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.20 to 0.63] — Odds Ratio of HbA1c <7% for Insulin Lispro 6 Day versus Insulin Aspart 6 Day

6. Other Pre Specified Outcome: Change From Baseline to 12 Weeks for Daily Insulin Dose (Total, Basal, and Bolus)
Time Frame: Baseline, endpoint for each 12-week treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units (U) of insulin
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 119 | 115
Units (U) of insulin
  Total Insulin Dose | 5.21 (8.94) | 4.97 (7.57)
  Basal Insulin Dose | 2.34 (3.51) | 1.91 (3.80)
  Bolus Insulin Dose (N=112, 112) | 2.19 (5.58) | 1.80 (4.70)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 0.595, Crossover Model — P-value for Total Insulin Dose computed using Crossover model: Variable = Treatment + Sequence + Period + Baseline Insulin Total Dose
Statistical Analysis 2: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 0.506, Crossover Model — P-value for Basal Insulin Dose computed using Crossover model: Variable = Treatment + Sequence + Period + Baseline Insulin Basal Dose
Statistical Analysis 3: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 0.790, Crossover Model — P-value for Bolus Insulin Dose computed using Crossover model: Variable = Treatment + Sequence + Period + Baseline Insulin Bolus Dose

7. Other Pre Specified Outcome: Percentage of Participants Having a Hyperglycemic Episode
Description: A hyperglycemic episode was defined as an event with (1) a measured blood glucose concentration >250 milligrams per deciliter (mg/dL) (13.9 millimoles per liter [mmol/L]) and ≥3 hours after eating, or (2) a measured blood glucose concentration >300 mg/dL (16.7 mmol/L) and <3 hours after eating
Time Frame: Days 1-6 for each reservoir cycle throughout each 12-week treatment period
Population: All randomized participants who received at least one dose of study drug. Participants included in hyperglycemia analyses are only those for whom data existed regarding hyperglycemia.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 124 | 124
percentage of participants | 97.6 | 98.4

8. Other Pre Specified Outcome: Hyperglycemic Episode Rate Per 30 Days
Description: Hyperglycemia was defined as an episode with (1) a measured blood glucose concentration >250 milligrams per deciliter [mg/dL] (13.9 millimoles per liter [mmol/L]) and ≥3 hours after eating, or (2) a measured blood glucose concentration >300 mg/dL (16.7 mmol/L) and <3 hours after eating. Rate is presented as the number of hyperglycemic episodes adjusted for 30 days.
Time Frame: Days 1-6 for each reservoir cycle throughout each 12-week treatment period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hyperglycemic episodes per 30 days
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 124 | 124
hyperglycemic episodes per 30 days | 15.47 (9.25) | 14.23 (10.19)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 0.059, negative binomial test; P-value computed using a negative binomial test including factors for treatment, period and sequence

9. Other Pre Specified Outcome: Percentage of Participants With Pump Complications
Description: Overall pump complications are defined as any combination of the following, reported by the participant: tubing clogged, tubing kinked, tubing disconnect, tubing pulled out, blood in tubing, too much heat, too much cold, empty reservoir, low battery, occlusion alarm, no delivery alarm, skin abscess at site, excessive redness at site, swelling (not nodule) at site, bleeding at site, bruising at site, reservoir change (infusion set change reason only), and other. When either a reservoir change or an infusion set change was reported, participants were questioned whether the change occurred early (prior to 6 days). If he/she responded 'yes', then the reported change was recorded as a premature change.
Time Frame: Days 1-6 for each reservoir cycle throughout each 12-week treatment period
Population: All randomized participants who completed at least one post-randomization visit. Participants included in pump complication analyses are only those for whom data existed regarding pump complications.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 127 | 127
percentage of participants
  Pump Complication: Premature Reservoir Change | 42.5 | 44.1
  Pump Complication: Premature Infusion Set Change | 74.8 | 70.9
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 1.00, Gart's Test — P-value for overall pump complications associated with a premature reservoir change computed using Gart's Test. Participants represented in both treatment groups and with non-missing incidence value in each treatment period are used
Statistical Analysis 2: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 0.472, Gart's Test — P-value for overall pump complications associated with a premature infusion set change computed using Gart's Test. Participants represented in both treatment groups and with non-missing incidence value in each treatment period are used

10. Other Pre Specified Outcome: Pump Complications Rate Per 30 Days
Description: Overall pump complications are defined as any combination of the following reported by the participant: tubing clogged, tubing kinked, tubing disconnect, tubing pulled out, blood in tubing, too much heat, too much cold, empty reservoir, low battery, occlusion alarm, no delivery alarm, skin abscess at site, excessive redness at site, swelling (not nodule) at site, bleeding at site, bruising at site, reservoir change (infusion set change reason only), and other. When either a reservoir change or an infusion set change was reported, participants were questioned whether the change occurred early (prior to 6 days). If he/she responded 'yes', then the reported change was recorded as a premature change.
Time Frame: Days 1-6 for each reservoir cycle throughout each 12-week treatment period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pump complications per 30 days
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 127 | 127
pump complications per 30 days
  Pump Complication: Premature Reservoir Change | 0.42 (0.93) | 0.45 (1.03)
  Pump Complication: Premature Infusion Set Change | 1.01 (1.41) | 1.10 (1.47)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 0.383, negative binomial test — P-value for Premature Reservoir Change computed using negative binomial test including factors for treatment, period and sequence
Statistical Analysis 2: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 0.499, negative binomial test — P-value for Premature Infusion Set Change computed using negative binomial test including factors for treatment, period and sequence

11. Other Pre Specified Outcome: Percentage of Participants Having a Hypoglycemic Episode
Description: A Documented Hypoglycemic Episode is defined as an event which is associated with a documented blood glucose (BG) concentration of <= 70 mg/dL (3.9 mmol/L).
  All Reported Hypoglycemic Episodes are defined as an event which is associated with
  1. reported signs and symptoms of hypoglycemia, and/or
  2. a documented blood glucose (BG) concentration of <= 70 mg/dL (3.9 mmol/L)
Time Frame: All days for each reservoir cycle throughout each 12-week treatment period
Population: All randomized participants who received at least one dose of study drug. Participants included in hypoglycemia analyses are only those for whom data existed regarding hypoglycemia.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 127 | 127
percentage of participants
  Documented Hypoglycemic Episodes | 91.3 | 93.7
  All Reported Hypoglycemic Episodes | 99.2 | 99.2
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 1.00, Gart's Test — The p-value is for the Documented Hypoglycemic Episodes category treatment arm comparison. The p-value for the All Reported Hypoglycemic Episodes category could not be generated using Gart's Test; Participants represented in both treatment groups, and with non-missing incidence value in each treatment period, were used for p-value calculation

12. Other Pre Specified Outcome: Hypoglycemic Episode Rate Per 30 Days
Description: All Reported Hypoglycemic Episodes are defined as an event which is associated with
  1. reported signs and symptoms of hypoglycemia, and/or
  2. a documented blood glucose (BG) concentration of <= 70 mg/dL (3.9 mmol/L)
Time Frame: All days for each reservoir cycle throughout each 12-week treatment period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hypoglycemic episodes per 30 days
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 127 | 127
hypoglycemic episodes per 30 days | 16.94 (10.69) | 18.90 (11.58)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p < 0.001, Negative Binomial Test; P-value computed using a negative binomial test including factors for treatment, period and sequence

13. Other Pre Specified Outcome: Change From Baseline to 12 Week Endpoint for Each Treatment in Weight
Time Frame: Baseline, endpoint for each 12-week treatment period
Population: All randomized participants who received at least one dose of study drug and had both baseline and post-baseline weight measurements for the respective treatment period.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 126 | 123
kilograms (kg) | -0.04 (2.25) | 0.56 (2.15)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p < 0.001, Crossover Model; P-value computed using crossover model. Response = treatment + sequence + period + baseline body weight

14. Other Pre Specified Outcome: Change From Baseline to 12 Weeks Endpoint for Each Treatment in Blood Pressure
Time Frame: Baseline, endpoint for each 12-week treatment period
Population: All randomized participants who received at least one dose of study drug and had both baseline and post-baseline blood pressure measurements for the respective treatment period.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Number analyzed (Participants) | 126 | 121
millimeters of mercury (mmHg)
  Systolic Blood Pressure (SBP) | -2.25 (14.71) | -1.36 (12.12)
  Diastolic Blood Pressure (DBP) | -1.61 (10.36) | -1.57 (9.13)
Statistical Analysis 1: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 0.147, Crossover Model — P-value for the Systolic Blood Pressure (SBP) computed using crossover model. Response = treatment + sequence + period + baseline systolic blood pressure
Statistical Analysis 2: Comparison: Insulin Lispro 6D vs Insulin Aspart 6D; Test type: Superiority or Other; p = 0.894, Crossover Model — P-value for Diastolic Blood Pressure (DBP) computed using crossover model. Response = treatment + sequence + period + baseline diastolic blood pressure

ADVERSE EVENTS:
Arm/Group | Insulin Lispro 6D | Insulin Aspart 6D
Serious Adverse Events (participants affected / at risk) | 3/127 | 7/127
Other Adverse Events (participants affected / at risk) | 34/127 | 31/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro 6D (N=127) | Insulin Aspart 6D (N=127)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (8) — These events were severe hypoglycemic events.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro 6D (N=127) | Insulin Aspart 6D (N=127)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Device occlusion (General disorders) | 1 (2) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 10 (10) | 6 (6)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Uterine infection (Infections and infestations) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Atherectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Injection (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Input to primary endpoint measurements (SMBG) contained approximately 40% missing data. Several analyses to account for missing data were conducted and results from these additional analyses were consistent with results from the original analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days